CLINICAL TRIAL: NCT05819710
Title: A Study to Investigate the Next-day Residual Effects of TS-142 in Healthy Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TS142-305
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2023-04

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — TS-142; zopiclone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 5 mg of TS-142 (Experimental): Low dose of TS-142
  Interventions: Drug: TS-142
- 10 mg of TS-142 (Experimental): High dose of TS-142
  Interventions: Drug: TS-142
- 7.5 mg of Zopiclone (Experimental): Comparator.
  Interventions: Drug: Zopiclone
- Placebo (Experimental): Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TS-142 — Single dose of 5 mg of TS-142
  Arms: 5 mg of TS-142
Drug: TS-142 — Single-dose of 10 mg of TS-142
  Arms: 10 mg of TS-142
Drug: Zopiclone — Single-dose of 7.5 mg of zopiclone
  Arms: 7.5 mg of Zopiclone
Drug: Placebo — Single-dose of placebo
  Arms: Placebo

SUMMARY:
This is a study to investigate the next-day residual effects of a single bedtime dosing of 5 mg and 10 mg of TS-142 in Japanese healthy elderly participants in double-blind manner.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are Japanese male or female aged 65 years or older at the time of obtaining informed consent
2. Subjects with a body Mass Index (BMI) from 18.5 to less than 25.0 and a body weight of 40.0 kg or over at the screening test
3. Subjects who are judged by the principal investigators or subinvestigators as an eligible for the clinical trial participation based on the results of tests conducted in the screening, VISIT 1 and prior to the administration of the investigational drug.

Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

1. Subjects who are judged to have any disease by the principal investigator or sub-investigator and are not considered healthy
2. Subjects who have any unsuitable medical histories for participation in this clinical trial, including respiratory, cardiovascular, gastrointestinal, hepatic, renal, urological, endocrinological, metabolic, hematologic, immunologic, dermatological, neurological, or psychiatric diseases
3. Subjects who have any medical histories including sleep-associated symptoms, narcolepsy-like symptoms, suicidal ideation, or suicidal attempts.

Other protocol defined exclusion criteria could apply.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
RMS of COP in eye-open condition | 8 hour postdose
  the area of the circle whose radius is the root mean square (RMS) value of center of pressure (COP) calculated by the stabilometer in eye-open condition

SECONDARY OUTCOMES:
RMS of COP in eye-closed condition | 8 hour postdose
  the area of the circle whose radius is the root mean square (RMS) value of center of pressure (COP) calculated by the stabilometer in eye-closed condition
Trajectory of COP in eye-open condition | 8 hour postdose
  the length of the total trajectory of center of pressure (COP) calculated by the stabilometer in eye-open condition
Trajectory of COP in eye-closed condition | 8 hour postdose
  the length of the total trajectory of center of pressure (COP) calculated by the stabilometer in eye-closed condition

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No